CLINICAL TRIAL: NCT02570451
Title: Preoperative Cognitive Screening of Surgical Patients 65 Years of Age or Older: Feasibility of Routine Screening and Utility for Predicting Morbidity
Brief Title: Preoperative Cognitive Screening of Surgical Patients 65 Years of Age or Older
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Anesthesia Patient Safety Foundation (Other)
Responsible Party: Principal Investigator, Gregory J. Crosby, M.D., Physician, Brigham and Women's Hospital
Other Study IDs: 2013P001214B
Record Dates: First submitted 2015-09-02; First posted 2015-10-07 (Estimated); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Mild Cognitive Impairment
Keywords: cognitive impairment; post surgical outcomes; elective joint replacement surgery
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Mental Status and Dementia Tests; Hand Strength

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- undergoing any elective SDA surgical procedure: 500 patients Patient Survey Independent Activities of Daily Living Score Sheet Geriatric Depression Scale Short Form Activities of Daily Living Score Sheet Grip Strength Mini Cog RAND 36-Item Short Form Health Survey Confusion Assessment Method (CAM)
  Interventions: Other: Patient Survey; Other: Mini Cog; Other: Independent Activities of Daily Living Score Sheet; Other: Activities of Daily Living Score Sheet; Other: Geriatric Depression Scale Short Form; Other: Confusion Assessment Method (CAM); Other: RAND 36-Item Short Form Health Survey; Other: Grip Strength
- scheduled for elective joint replacement surgery: Patient Survey Independent Activities of Daily Living Score Sheet Geriatric Depression Scale Short Form 211 patients Activities of Daily Living Score Sheet Grip Strength Mini Cog RAND 36-Item Short Form Health Survey Confusion Assessment Method (CAM)
  Interventions: Other: Patient Survey; Other: Mini Cog; Other: Independent Activities of Daily Living Score Sheet; Other: Activities of Daily Living Score Sheet; Other: Geriatric Depression Scale Short Form; Other: Confusion Assessment Method (CAM); Other: RAND 36-Item Short Form Health Survey; Other: Grip Strength

INTERVENTIONS:
Other: Patient Survey — This survey will assess patients' perspective about the importance of preoperative cognitive screening, information about living situation, information about who accompanied them to the preoperative visit, and level of perceived stress.
Other: Mini Cog — The MiniCog is a simple cognitive screening tool that takes just 2-4 min to complete and has little or no education, language, or race bias. This is a well-validated tool to assess mild cognitive impairment.
Other: Independent Activities of Daily Living Score Sheet — Questionnaire used to measure self-reported functional status for instrumental activities of daily living using standardized scales
  Other Names: IADLs
Other: Activities of Daily Living Score Sheet — Questionnaire used to measure self-reported functional status for basic activities of daily living using standardized scores
  Other Names: ADLs
Other: Geriatric Depression Scale Short Form — Questionnaire used to measure self-reported mood
  Other Names: GDS
Other: Confusion Assessment Method (CAM) — This well-validated measure of post-operative delirium will be utilized up to 3 days after surgery
Other: RAND 36-Item Short Form Health Survey — This measure is a generic, coherent, and easily administered health survey used to assess self-reported quality of life
Other: Grip Strength — Measured using the JAMAR dynamometer

SUMMARY:
The overall objectives of this study are to improve outcomes of surgical patients 65 years of age or older through risk stratification based on preoperative screening of cognition / mental function. Aim 1 is to determine the prevalence of cognitive impairment among patients 65 years of age or older presenting for elective joint replacement surgery by structured cognitive screening versus standard practice. Aim 2 is to ascertain whether preoperative cognitive impairment in patients 65 years of age or older undergoing elective joint replacement surgery is an independent predictor of adverse postoperative events and/or mortality. Aim 3 is to implement routine structured preoperative cognitive screening of patients 65 years of age or older undergoing elective surgical procedures in a busy preoperative clinic.

DETAILED DESCRIPTION:
This will be a prospective, single-center observational study of patients 65 years of age or older undergoing elective surgical procedures. Phase 1 (Aims 1 and 2), will examine the prevalence of preoperative cognitive impairment and its relationship to postoperative outcome. In Phase 2 (Aim 3), will implement routine structured cognitive screening in a busy surgical preadmission evaluation center and confirm its utility for predicting adverse perioperative outcomes in elders.

For Phase 1, 211 randomly selected patients 65 years of age or older of either gender will be enrolled presenting to the Brigham and Women's Hospital Weiner Center for Preoperative Evaluation (CPE) scheduled for elective joint replacement surgery. The Brigham and Women's Hospital performs more than 600 joint replacement procedures each year in patients 65 years of age or older. This is the age range where cognitive impairment becomes prevalent and postoperative cognitive and non-cognitive morbidity is common. Exclusion criteria will be patients diagnosed with dementia or cognitive impairment; scheduled for a procedure affecting the brain or cerebrovasculature (i.e. intracranial neurosurgery, carotid endarterectomy, cardiac surgery); planned to go to an ICU postoperatively; with uncorrected vision or hearing impairment (who cannot see the pictures or read or hear instructions); unable to use their dominant hand (limited ability to draw); and/or unable to speak, read or understand English. The investigators will use the CPE computerized scheduling system, which is updated continuously in real time and captures relevant information such as age and procedure to identify potential subjects. When patients check in with the receptionist for their appointment they will be notified that they may be eligible to participate in a study involving patients 65 years of age or older. The receptionist will then provide them with a brochure about the study that includes information about the purpose of the study, the risks to the patient, and potential benefits to society. The patient will then be asked if they are willing to speak with one of the study investigators and only those patients that agree to speak with a study investigator will be approached. A member of the study team will then contact the patient and verify that they satisfy the inclusion criteria and discuss the goals and risks of the study and ask them to participate. After all questions have been answered and the patient has had an opportunity to read the consent form, written consent will be obtained. After obtaining consent the patient will be interviewed by a member of the study team to obtain information about their years of education and self-reported functional status according to standardized scales for basic and instrumental activities of daily living (ADLs and IADLs, respectively). Grip strength as an index of frailty and mood assessed with the Geriatric Depression Scale-Short (GDS). An investigator will also administer a survey to assess the patient's perspective about the importance of preoperative cognitive screening. Information about ASA physical status, medications, and Charlson comorbidity index will be extracted subsequently from the patient's electronic medical record and patient interview. The patient will then be administered the MiniCog a simple cognitive screening tools that take just 2-4 min to complete and has little or no education, language, or race bias. During this phase of the project, a trained study team member will administer the test in the quiet of the evaluation room. The practitioner conducting the actual preoperative evaluation will be blinded to the cognitive test results and will complete a questionnaire about the patient's cognitive status based on their interactions during the visit. A trained, blinded member of the study team will score the test. Discharge to place other than home will be used as the primary outcome to determine the relationship between pre-existing cognitive impairment and patient outcome (Aim 2). As a secondary outcome delirium will be assessed once per day on postoperative days 1, 2, and 3 by a member of the study team using the Confusion Assessment Method (CAM) a well-validated measure of delirium in surgical patients. Other secondary outcomes that will be evaluated will include the use of restraints, hospital length of stay (LOS), complications (including in-hospital falls), 30 d readmission rate, and 30 d, 6 month, 1 year and 5 year mortality. Data will be extracted from the medical record and the BWH Balanced Scorecard. Phase 2 will examine the feasibility of implementing routine structured cognitive screening for elective surgical procedures into a busy preoperative evaluation center. 500 patients will be enrolled according to the criteria outlined above and ask CPE practitioners to administer the structured cognitive screen to all patient ≥ 65 years of age scheduled for a surgical procedure as part of their routine preoperative evaluation. A study team member will train the CPE staff in administration of the MiniCog prior to beginning this phase of the study; the test will be administered as part of the routine CPE visit. Outcome measures will be rate of successful testing (a score-able test), and impact of testing on patient flow. The latter will be obtained by extracting and comparing data from the CPE's computerized patient flow tracking system on time spent with a provider in a preoperative evaluation room and total duration of the CPE visit (check-in time to departure time) between enrolled subjects and age and procedure matched patients seen in the CPE the previous year.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older
* scheduled for elective joint replacement surgery

Exclusion Criteria:

* Known diagnosis of dementia or cognitive impairment
* Uncorrected vision or hearing impairment
* Unable to use dominant hand to write
* Unable to speak, read, or understand English

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients 65 years or older in the Weiner Center for Preoperative Evaluation presenting for elective joint replacement surgery
Sampling Method: Non-Probability Sample
Enrollment: 711 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Discharge location (defined home vs. other than home) on day of patient discharge from hospital | up to 30 days after surgery
  On the day the patient is discharged from the hospital, the discharge location (home vs. other than home) will be recorded

SECONDARY OUTCOMES:
Patient score on the confusion assessment method postoperative days 1-3 | up to 3 days after surgery
  Delirium will be measured using the Confusion Assessment Method (CAM) by a member of the study team on postoperative days 1, 2 and 3
Number of newly diagnosed health complications following surgery | up to 30 days after surgery
  Number of newly diagnosed health complications will be recorded up to 30 days after surgery including: Myocardial Infarction, CHF, Cardiac Arrest, Arrythmia, Pneumonia, PE, Reintubation, Stroke, Delirium, Coma>24h, Postoperative deep wound infection, Superficial wound infection, Sepsis, Renal Failure, UTI, Reoperation, DVT, ICU admission
Readmission Rate | up to 30 days after surgery
  Whether or not patients are readmitted to the hospital within 30 days of discharge after surgery
Emergency Room Admit | up to 30 days after surgery
  Whether or not patients are admitted to the ER within 30 days of discharge after surgery
Mortality | up to 5 years after surgery
  Patient mortality within 30 days of being discharged from the hospital post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Deborah J Culley, M.D., Principal Investigator — Brigham and Women's Anesthesiology Department
Locations (1):
- Weiner Center for Preoperative Evaluation, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided